CLINICAL TRIAL: NCT04723355
Title: A Comparative Study of the Findings of Dynamic Electrocardiography (Holter System) Using the an Innovative 3-lead Wireless Water Resistant Device and a Conventional Device
Brief Title: A Comparative Study of an Innovative 3-lead Wireless Water Resistant Holter System and a Conventional Holter System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other); Quoretech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 40422220.1.0000.5462
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Holter device (Experimental): In this single arm of the study, the participant will use 2 Holter systems simultaneously for 24 hours, an innovative 3-lead wireless water resistant device and a conventional device.
  Interventions: Device: An innovative 3-lead wireless water resistant Holter device; Device: A conventional device

INTERVENTIONS:
Device: An innovative 3-lead wireless water resistant Holter device — The participant will use the innovative 3-lead wireless water resistant Holter device simultaneously with the conventional Holter device for 24 hours.
Device: A conventional device — The participant will use the innovative 3-lead wireless water resistant Holter device simultaneously with the conventional Holter device for 24 hours.

SUMMARY:
Holter monitoring is one of the most widely used diagnostic methods to detect cardiac arrhythmias. Newer Holter monitors may provide some advantages over the more traditional ones. This study will compare the findings of a Holter exam using an innovative 3-lead wireless water resistant device with a conventional device.

DETAILED DESCRIPTION:
The 24-hour ambulatory electrocardiography, commonly known as Holter monitoring, is a diagnostic method to correlate clinical symptoms with cardiac arrhythmias. The Holter monitor records electrical signals from the heart using electrodes attached to the chest, which are connected via cables to a digital recorder. In addition to the device to record the cardiac electrical signals, the Holter system also has a software for review and analysis of the record. The software of the Holter system has an integrated automatic analysis process to detect different sorts of heart beats, rhythms, etc, which are then validated by a technician and a physician. The success of the automatic analysis depends of the quality of the captured electrical signals, which are dependent on the appropriate attachment of the electrodes/cables to the patient body. Therefore, inappropriately attached electrodes/cables can result in electromagnetic disturbance that can interfere with the ECG signal, resulting in a very noisy record that is hard to be analysed.

Newer Holter systems that eliminate the cables and attach the recorder directly to the electrodes positioned in the patient´s chest might reduce the electromagnetic disturbance in the ECG signal capture and, therefore, improve the quality of the exam.

This study will compare the findings of a Holter exam using an innovative 3-lead wireless water resistant device with a conventional device.

ELIGIBILITY:
Inclusion Criteria:

* Any individual who has an indication of 24 hours Holter monitoring and is referred to the arrhythmia clinic of the Instituto Dante Pazzanese de Cardiologia

Exclusion Criteria:

* Refusal to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karla Santo, PhD, Study Director — Hospital Israelita Albert Einstein
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared upon review of a request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals attending the study inclusion criteria were consecutively approached to participate in the study between 26 January 2021 and 16 November 2021 at the arrhythmia clinic of the Instituto Dante Pazzanese de Cardiologia in Sao Paulo, Brazil
Period: Overall Study
Arm/Group | Holter Device
Started | 231
Completed | 179
Not Completed | 52
Not completed — Issues with leads off, substantial ECG signal artefacts, and ECG data upload errors | 50
Not completed — Errors in the informed consent form | 2

BASELINE CHARACTERISTICS:
Arm/Group | Holter Device
Number analyzed (Participants) | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 113
  Race: Mixed | 35
  Race: Black | 29
  Race: Asian | 2
Region of Enrollment [Number; unit: participants]
  Brazil | 179
Marital status [Count of Participants; unit: Participants]
  Married | 115
  Single | 30
  Divorced | 19
  Widowed | 15
Level of education [Count of Participants; unit: Participants]
  Illiterate | 1
  Incomplete primary school | 21
  Complete primary school | 61
  Complete secondary school | 57
  Complete technical school | 2
  Incomplete undergraduate school | 9
  Complete undergraduate school | 26
  Complete postgraduate school | 2
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (4.8)
Hypertension [Count of Participants; unit: Participants]
  Yes | 123
  No | 48
  Missing | 8
Diabetes [Count of Participants; unit: Participants]
  Yes | 39
  No | 130
  Did not know | 2
  Missing | 8
Heart failure [Count of Participants; unit: Participants]
  Yes | 86
  No | 81
  Did not know | 2
  Missing | 10
Previous myocardial infarction [Count of Participants; unit: Participants]
  Yes | 42
  No | 128
  Did not know | 1
  Missing | 8
Previous stroke [Count of Participants; unit: Participants]
  Yes | 36
  No | 92
  Did not know | 1
  Missing | 50
Hypothyroidism [Count of Participants; unit: Participants]
  Yes | 20
  No | 106
  Did not know | 3
  Missing | 50
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants]
  Yes | 11
  No | 117
  Did not know | 1
  Missing | 50

OUTCOME MEASURES:

1. Primary Outcome: Detection of Cardiac Arrhythmias
Description: Number of patients with cardiac arrhythmias detected in both Holter monitors, including a) atrial fibrillation or atrial flutter; b) supraventricular tachycardia (any tachycardia with ≥ 3 beats arising outside the sinus node and above the His-Purkinje bifurcation, including atrial tachycardia, atrioventricular nodal reentry tachycardia, junctional tachycardia and accessory pathway reentry tachycardia, except atrial fibrillation and atrial flutter); c) ventricular tachycardia (any tachycardia with ≥ 3 beats arising from the ventricles, except polymorphic ventricular tachycardia or ventricular fibrillation); d) polymorphic ventricular tachycardia or ventricular fibrillation; e) atrioventricular (AV) block (high-degree AV block, in which there is an interruption in the transmission of a heart beat from the atria to the ventricles, including those classified as 2nd degree AV block Mobitz type I and II, AV block 2:1 or complete AV block); or f) heart beat pauses (≥ 2,5 seconds)
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Device
Number analyzed (Participants) | 179
Participants
  Innovative 3-lead Wireless Water Resistant Holter System | 107
  Conventional Holter System | 104
Statistical Analysis 1: Comparison: Holter Device; The comparison of the two Holter monitoring devices was analyzed in terms of the accuracy of the Innovative 3-lead Wireless Water Resistant Holter System in detecting the arrhythmias compared to the Conventional Holter System as the gold standard; Test type: Non-Inferiority — In the sample size calculations, we assumed that the innovative 3-lead wireless water resistant Holter System would have a concordance in the diagnosis of arrhythmia compared to the conventional Holter device similar to a previous study that compared a patch to the conventional Holter device. With this assumption, a total sample of 182 participants would have 80% power to demonstrate an accuracy of at least 85% with a significance level of 2.5% (the 95% CI lower limit should be above 85%); Accuracy = 0.87, 95% CI 2-sided [0.81 to 0.92]
Statistical Analysis 2: Comparison: Holter Device; Other measures of diagnostic accuracy, including the sensitivity, specificity, positive and negative predictive values were also analyzed; Test type: Other; Sensitivity = 0.90, 95% CI 2-sided [0.83 to 0.95]
Statistical Analysis 3: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Specificity = 0.83, 95% CI 2-sided [0.72 to 0.90]
Statistical Analysis 4: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Positive predictive value = 0.88, 95% CI 2-sided [0.80 to 0.93]
Statistical Analysis 5: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Negative predictive value = 0.86, 95% CI 2-sided [0.76 to 0.93]
Statistical Analysis 6: Comparison: Holter Device; We also did an additional analysis to further evaluate the concordance between both Holter monitoring devices using the Cohen´s Kappa coefficient; Test type: Other; Cohen Kappa coefficient = 0.74
Statistical Analysis 7: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Positive likelihood ratio = 5.21, 95% CI 2-sided [3.17 to 8.58]
Statistical Analysis 8: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Negative likelihood ratio = 0.12, 95% CI 2-sided [0.06 to 0.21]

2. Secondary Outcome: Detection of Atrial Fibrillation or Atrial Flutter
Description: Number of patients with atrial fibrillation or atrial flutter detected in both Holter monitors
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Device
Number analyzed (Participants) | 179
Participants
  Innovative 3-lead Wireless Water Resistant Holter System | 23
  Conventional Holter System | 22
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 1, analysis 1]; Test type: Other; Accuracy = 0.99, 95% CI 2-sided [0.97 to 1.00]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Sensitivity = 1.00, 95% CI 2-sided [0.85 to 1.00]
Statistical Analysis 3: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Specificity = 0.99, 95% CI 2-sided [0.97 to 1.00]
Statistical Analysis 4: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Positive predictive value = 0.96, 95% CI 2-sided [0.78 to 1.00]
Statistical Analysis 5: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Negative predictive value = 1.00, 95% CI 2-sided [0.98 to 1.00]
Statistical Analysis 6: Comparison: Holter Device; [analysis description as in outcome 1, analysis 6]; Test type: Other; Cohen Kappa coefficient = 0.97
Statistical Analysis 7: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Positive likelihood ratio = 157, 95% CI 2-sided [22.25 to 1107.61]
Statistical Analysis 8: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Negative likelihood ratio = 0.0, 95% CI 2-sided [0 to 0]

3. Secondary Outcome: Detection of Supraventricular Tachycardia
Description: Number of patients with supraventricular tachycardia (any tachycardia with ≥ 3 beats arising outside the sinus node and above the His-Purkinje bifurcation, including atrial tachycardia, atrioventricular nodal reentry tachycardia, junctional tachycardia and accessory pathway reentry tachycardia, except atrial fibrillation and atrial flutter) detected in both Holter monitors
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Device
Number analyzed (Participants) | 179
Participants
  Innovative 3-lead Wireless Water Resistant Holter System | 71
  Conventional Holter System | 71
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 1, analysis 1]; Test type: Other; Accuracy = 0.85, 95% CI 2-sided [0.79 to 0.90]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Sensitivity = 0.82, 95% CI 2-sided [0.71 to 0.90]
Statistical Analysis 3: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Specificity = 0.88, 95% CI 2-sided [0.80 to 0.93]
Statistical Analysis 4: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Positive predictive value = 0.82, 95% CI 2-sided [0.71 to 0.90]
Statistical Analysis 5: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Negative predictive value = 0.88, 95% CI 2-sided [0.80 to 0.93]
Statistical Analysis 6: Comparison: Holter Device; [analysis description as in outcome 1, analysis 6]; Test type: Other; Cohen Kappa coefficient = 0.70
Statistical Analysis 7: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Positive likelihood ratio = 6.79, 95% CI 2-sided [4.03 to 11.43]
Statistical Analysis 8: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Negative likelihood ratio = 0.21, 95% CI 2-sided [0.13 to 0.34]

4. Secondary Outcome: Detection of Ventricular Tachycardia
Description: Number of patients with ventricular tachycardia (any tachycardia with ≥ 3 beats arising from the ventricles, except polymorphic ventricular tachycardia or ventricular fibrillation) detected in both Holter monitors
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Device
Number analyzed (Participants) | 179
Participants
  Innovative 3-lead Wireless Water Resistant Holter System | 26
  Conventional Holter System | 23
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 1, analysis 1]; Test type: Other; Accuracy = 0.93, 95% CI 2-sided [0.88 to 0.96]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Sensitivity = 0.78, 95% CI 2-sided [0.56 to 0.93]
Statistical Analysis 3: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Specificity = 0.95, 95% CI 2-sided [0.90 to 0.98]
Statistical Analysis 4: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Positive predictive value = 0.69, 95% CI 2-sided [0.48 to 0.86]
Statistical Analysis 5: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Negative predictive value = 0.97, 95% CI 2-sided [0.93 to 0.99]
Statistical Analysis 6: Comparison: Holter Device; [analysis description as in outcome 1, analysis 6]; Test type: Other; Cohen Kappa coefficient = 0.69
Statistical Analysis 7: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Positive likelihood ratio = 15.26, 95% CI 2-sided [7.51 to 30.99]
Statistical Analysis 8: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Negative likelihood ratio = 0.23, 95% CI 2-sided [0.11 to 0.50]

5. Secondary Outcome: Detection of Polymorphic Ventricular Tachycardia or Ventricular Fibrillation
Description: Number of patients with polymorphic ventricular tachycardia or ventricular fibrillation detected in both Holter monitors
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Device
Number analyzed (Participants) | 179
Participants
  Innovative 3-lead Wireless Water Resistant Holter System | 14
  Conventional Holter System | 12
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 1, analysis 1]; Test type: Other; Accuracy = 0.93, 95% CI 2-sided [0.89 to 0.96]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Sensitivity = 0.58, 95% CI 2-sided [0.28 to 0.85]
Statistical Analysis 3: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Specificity = 0.96, 95% CI 2-sided [0.92 to 0.98]
Statistical Analysis 4: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Positive predictive value = 0.50, 95% CI 2-sided [0.23 to 0.77]
Statistical Analysis 5: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Negative predictive value = 0.97, 95% CI 2-sided [0.93 to 0.99]
Statistical Analysis 6: Comparison: Holter Device; [analysis description as in outcome 1, analysis 6]; Test type: Other; Cohen Kappa coefficient = 0.77
Statistical Analysis 7: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Positive likelihood ratio = 13.92, 95% CI 2-sided [5.84 to 33.17]
Statistical Analysis 8: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Negative likelihood ratio = 0.43, 95% CI 2-sided [0.22 to 0.85]

6. Secondary Outcome: Detection of Atrioventricular Block
Description: Number of patients with atrioventricular block (high-degree AV block, in which there is an interruption in the transmission of a heart beat from the atria to the ventricles, including those classified as 2nd degree AV block Mobitz type I and II, AV block 2:1 or complete AV block) detected in both Holter monitors
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Device
Number analyzed (Participants) | 179
Participants
  Innovative 3-lead Wireless Water Resistant Holter System | 5
  Conventional Holter System | 4
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 1, analysis 1]; Test type: Other; Accuracy = 0.98, 95% CI 2-sided [0.95 to 1.00]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Sensitivity = 0.75, 95% CI 2-sided [0.19 to 0.99]
Statistical Analysis 3: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Specificity = 0.99, 95% CI 2-sided [0.96 to 1.00]
Statistical Analysis 4: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Positive predictive value = 0.60, 95% CI 2-sided [0.15 to 0.95]
Statistical Analysis 5: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Negative predictive value = 0.99, 95% CI 2-sided [0.97 to 1.00]
Statistical Analysis 6: Comparison: Holter Device; [analysis description as in outcome 1, analysis 6]; Test type: Other; Cohen Kappa coefficient = 0.66
Statistical Analysis 7: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Positive likelihood ratio = 65.63, 95% CI 2-sided [14.80 to 291.07]
Statistical Analysis 8: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Negative likelihood ratio = 0.25, 95% CI 2-sided [0.05 to 1.38]

7. Secondary Outcome: Detection of Heart Beat Pauses
Description: Number of patients with heart beat pauses ≥ 2.5 seconds detected in both Holter monitors
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Device
Number analyzed (Participants) | 179
Participants
  Innovative 3-lead Wireless Water Resistant Holter System | 7
  Conventional Holter System | 11
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 1, analysis 1]; Test type: Other; Accuracy = 0.98, 95% CI 2-sided [0.94 to 0.99]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Sensitivity = 0.64, 95% CI 2-sided [0.31 to 0.89]
Statistical Analysis 3: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Specificity = 1.00, 95% CI 2-sided [0.98 to 1.00]
Statistical Analysis 4: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Positive predictive value = 1.00, 95% CI 2-sided [0.59 to 1.00]
Statistical Analysis 5: Comparison: Holter Device; [analysis description as in outcome 1, analysis 2]; Test type: Other; Negative predictive value = 0.98, 95% CI 2-sided [0.94 to 0.99]
Statistical Analysis 6: Comparison: Holter Device; [analysis description as in outcome 1, analysis 6]; Test type: Other; Cohen Kappa coefficient = 0.77
Statistical Analysis 7: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; The positive likelihood ratio could not be calculated due to the value of zero in the denominator
Statistical Analysis 8: Comparison: Holter Device; Exploratory analyses of positive and negative likelihood ratios were also conducted; Test type: Other; Negative likelihood ratio = 0.36, 95% CI 2-sided [0.17 to 0.79]

8. Secondary Outcome: Duration of the Holter Exam
Description: Duration of the Holter exam in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Holter Device
Number analyzed (Participants) | 179
hours
  Innovative 3-lead Wireless Water Resistant Holter System | 21.79 (1.40)
  Conventional Holter System | 21.74 (1.95)

9. Secondary Outcome: Mean Heart Rate
Description: Mean heart rate measured in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Holter Device
Number analyzed (Participants) | 179
beats per minute
  Innovative 3-lead Wireless Water Resistant Holter System | 69.73 (12.10)
  Conventional Holter System | 70.67 (12.24)
Statistical Analysis 1: Comparison: Holter Device; The quantitative secondary outcomes were analyzed using Bland-Altman graphs as well as the Lin´s concordance correlation coefficient (CCC); Test type: Other; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-6.20 to 4.31]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Lin´s concordance correlation coeficient = 0.97, 95% CI 2-sided [0.96 to 0.98]

10. Secondary Outcome: Maximum Heart Rate
Description: Maximum heart rate measured in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Holter Device
Number analyzed (Participants) | 179
beats per minute
  Innovative 3-lead Wireless Water Resistant Holter System | 113.59 (23.17)
  Conventional Holter System | 116.30 (24.76)
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Mean Difference (Final Values) = -2.71, 95% CI 2-sided [-17.09 to 11.67]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Lin´s concordance correlation coeficient = 0.95, 95% CI 2-sided [0.93 to 0.96]

11. Secondary Outcome: Minimum Heart Rate
Description: Minimum heart rate measured in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Holter Device
Number analyzed (Participants) | 179
beats per minute
  Innovative 3-lead Wireless Water Resistant Holter System | 49.56 (9.83)
  Conventional Holter System | 49.17 (8.87)
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [-5.43 to 6.22]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Lin´s concordance correlation coeficient = 0.95, 95% CI 2-sided [0.93 to 0.96]

12. Secondary Outcome: Atrial Ectopic Heart Beats
Description: Total number of atrial ectopic heart beats measured in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: atrial ectopic heart beats in 24 hr
Arm/Group | Holter Device
Number analyzed (Participants) | 179
atrial ectopic heart beats in 24 hr
  Innovative 3-lead Wireless Water Resistant Holter System | 717.09 (2323.94)
  Conventional Holter System | 723.46 (2223.27)
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Mean Difference (Final Values) = -6.37, 95% CI 2-sided [-1391.46 to 1378.72]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Lin´s concordance correlation coeficient = 0.95, 95% CI 2-sided [0.94 to 0.96]

13. Secondary Outcome: Ventricular Ectopic Heart Beats
Description: Total number of ventricular ectopic heart beats measured in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ventricular ectopic heart beats in 24 hr
Arm/Group | Holter Device
Number analyzed (Participants) | 179
ventricular ectopic heart beats in 24 hr
  Innovative 3-lead Wireless Water Resistant Holter System | 1198.89 (2651.33)
  Conventional Holter System | 1187.85 (2696.69)
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Mean Difference (Final Values) = 11.04, 95% CI 2-sided [-2089.58 to 2111.65]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Lin´s concordance correlation coeficient = 0.92, 95% CI 2-sided [0.89 to 0.94]

14. Secondary Outcome: Episodes of Ventricular Tachycardia
Description: Total number of ventricular tachycardia episodes detected in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ventricular tachycardia episodes in 24hr
Arm/Group | Holter Device
Number analyzed (Participants) | 179
ventricular tachycardia episodes in 24hr
  Innovative 3-lead Wireless Water Resistant Holter System | 1.12 (6.29)
  Conventional Holter System | 1.24 (7.86)
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-5.45 to 5.20]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Lin´s concordance correlation coeficient = 0.93, 95% CI 2-sided [0.91 to 0.94]

15. Secondary Outcome: Episodes of Supraventricular Tachycardia
Description: Total number of supraventricular tachycardia episodes detected in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: supraventricular tachycardia episodes
Arm/Group | Holter Device
Number analyzed (Participants) | 179
supraventricular tachycardia episodes
  Innovative 3-lead Wireless Water Resistant Holter System | 5.71 (38.59)
  Conventional Holter System | 6.37 (41.10)
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-13.38 to 12.07]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Lin´s concordance correlation coeficient = 0.987, 95% CI 2-sided [0.98 to 0.99]

16. Secondary Outcome: Episodes of Heart Beat Pauses
Description: Total number of heart beat pauses ≥ 2.5 seconds detected in both Holter monitors
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: heart beat pauses in 24hr
Arm/Group | Holter Device
Number analyzed (Participants) | 179
heart beat pauses in 24hr
  Innovative 3-lead Wireless Water Resistant Holter System | 1.74 (12.13)
  Conventional Holter System | 1.84 (12.43)
Statistical Analysis 1: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.75 to 1.56]
Statistical Analysis 2: Comparison: Holter Device; [analysis description as in outcome 9, analysis 1]; Test type: Other; Lin´s concordance correlation coeficient = 0.9976, 95% CI 2-sided [0.997 to 0.998]

17. Secondary Outcome: Holter System Convenience of Use
Description: Number of Participants Reporting the convenience of use of the Holter systems
Time Frame: 24 hours
Population: Only 98 participants of the total of 179 responded the survey to assess the convenience of use of the Holter systems
Measure: Count of Participants; unit: Participants
Arm/Group | Holter Device
Number analyzed (Participants) | 98
Participants
  Innovative 3-lead Wireless Water Resistant Holter System | 54
  Conventional Holter System | 14
  No difference | 30
Statistical Analysis 1: Comparison: Holter Device; Test type: Superiority; p < 0.0001, Chi-squared; chi-squared test statistic = 23.529

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Holter Device
All-Cause Mortality (participants affected / at risk) | 0/179
Serious Adverse Events (participants affected / at risk) | 0/179
Other Adverse Events (participants affected / at risk) | 0/179

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It was agreed with the funding source that the trial results will be published in the Clinicaltrials.gov only.

DOCUMENTS (2):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT04723355/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT04723355/SAP_001.pdf